CLINICAL TRIAL: NCT06177158
Title: Efficacy of Oral Hygiene Instructions on Proinflammatory Cytokines Among Cigarette Smokers and Individuals Vaping Electronic Cigarettes During Plaque Induced Gingivitis (Clinical Trial)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Abdulrahman alauldin khazaal, B.D.S, University of Baghdad
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: vaping effect on biomarkers
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Electronic Cigarette Use; Plaque Induced Gingivitis
Keywords: smoking; Electronic Cigarette Use; Gingivitis
MeSH Terms: conditions — Vaping; Smoking; Gingivitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: lab technician and statistician will be masked
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- cigarette smoker with gingivitis. (Active Comparator): oral hygiene instructions
  Interventions: Behavioral: oral hygiene instructions
- electronic cigarette smoker with gingivitis. (Active Comparator): oral hygiene instructions
  Interventions: Behavioral: oral hygiene instructions
- non-smoker with gingivitis. (Active Comparator): oral hygiene instructions
  Interventions: Behavioral: oral hygiene instructions

INTERVENTIONS:
Behavioral: oral hygiene instructions — Standardized motivation and oral hygiene instructions regarding the tooth brushing will be demonstrated to all three groups using modified bass technique and a standardized brush, medium bristled brush with toothpaste, the patients will be instructed to brush their teeth for 2 minutes with a pea- size amount of dentifrice twice daily. For interdental cleaning aids each patient will be instructed to use the suitable methods regarding the space between teeth.
  clinically for each patient to ensure that the patients understood the instruction sessions. Before receiving oral hygiene instructions and motivation, the salivary sample will be collected and clinical periodontal parameters will be measured at a base line visit then, after 3 weeks, saliva will be collected and the same clinical measurements will be taken.

SUMMARY:
To evaluate the level of proinflammatory cytokines in individual vaping electronic cigarette in gingivitis patients.

Can vaping affects the proinflammatory cytokines level in diseased individuals?

Group I: cigarette smoker with gingivitis. Group II: electronic cigarette smoker with gingivitis. Group III: non-smoker with gingivitis.

participants will be asked to perform oral hygiene instructions.

measurement of inflammatory biomarkers MMP8 and MMP9 base line and after intervention will be done.

DETAILED DESCRIPTION:
Periodontal diseases are defined as an inflammatory process associated with bacterial activity and mediated by the host's immunologic response (Armitage, 1999; Tonetti et al., 2018). Gingivitis, a reversible form of periodontal disease, is initially characterized by gingival inflammation cause by bacterial colonization forming the biofilm (Armitage, 1999; Tonetti et al., 2018). Cigarette smoking is a classical risk factor for both periodontal and peri-implant tissue damage (Sgolastra et al., 2013). It has been shown that patients who smoke suffer from more severe forms of periodontitis (Javed et al., 2013).

Disease progression is directly related to the frequency of smoking, where heavy smokers show more severe forms of the disease compared to light smokers (Tonetti et al., 2018). Different studies categorize the frequency of smoking differently but according to one review, smoking less than 9 cigarettes per day is considered light, and more than 31 is considered heavy smoking (Johnson & Guthmiller, 2000). Smoking also impacts the response to periodontal treatment; smokers show only 50%-75% improvement in their clinical parameters after scaling and root planing compared to non-smokers (Tonetti et al., 2018).

Another study analyzed the effects of cigarette smoking on periodontal parameters and found significant increases in plaque index, pocket depth, and clinical attachment loss levels in cigarette smokers compared to non-smokers (Javed et al., 2017). It has been evidenced that tobacco smoking results in a proinflammatory effect by stimulating the secretion of specific cytokines and radical oxygen species (ROS) that play a role in the destruction of periodontal tissues (Katz et al., 2005) Electronic cigarettes (e-cigs) are battery-operated handheld devices, in which an e-liquid (contain ning nicotine and sometimes artificial flavors such as menthol, coffee, candy, butter and fruits) is heated by a heating element releasing a chemical-filled aerosol for inhalation (Sundar et al., 2016).

In the United States (U.S.), the use e-cigs is escalating predominantly in younger adults (Delnevo et al., 2015). Vaping without nicotine still proposes risks of exposure to the chemicals that are released in the heating process of the device, such as aluminum, copper, and lead (Gaur & Agnihotri, 2019). E-cigarettes also pose a hazard for traumatic injuries. Blast injuries caused by battery explosion are also an associated risk, mainly in countries where there is no regulation on the manufacture and safety of e-cigarettes (Kite et al., 2016).

Focusing on a correlation between oral health and vaping, a recent study showed that e-cigarette exposure-mediated carbonyl stress leads to increased levels of prostaglandin-E2 and cyclooxygenase-2 in human gingival epithelium compared to control (Lerner et al., 2015) Several studies analyzed the impact of vaping on periodontal parameters and found increased levels of plaque index, pocket depth, clinical attachment loss, and marginal bone loss in vaping groups compared to non-smokers (Al-Aali et al., 2018) Despite all the evidence that smoking can negatively affect the periodontal tissues, there is still little evidence about the impact of vaping(Figueredo et al., 2020).

So, the research question of current study will be: can vaping affect the level of proinflammatory cytokines in diseased samples.

Aim To evaluate the level of proinflammatory cytokines in individual vaping electronic cigarette in gingivitis patients.

Rationale Vaping can affect the periodontal health in many ways, a better understanding about the impact of vaping on periodontal health could pave the way to develop a better treatment plan for those patients.

Research Hypothesis

Null hypothesis: vaping has no effect on the proinflammatory cytokines level in diseased individuals.

Alternative hypothesis vaping affects the proinflammatory cytokines level in diseased individuals.

Methodology

Settings:

The study will be conducted at College of Dentistry/University of Baghdad / Iraq the study will be started at December 2023 till June 2024.

Adherence Printed follow-up schedule cards with reminder calls or messages will be utilized to remind the participants twice daily for brushing and using the intervention. Furthermore, the patient instructed to bring the container of mouth wash and interdental aids at the end point therapy.

Saliva collection and analysis Saliva will be collected as previously described before clinical examination (Zhang, Y et al, 2021). Participants will be asked to refrain from eating, drinking, or engaging in oral hygiene procedures for at least two hours prior saliva collection. Then, participants will rinse their mouths with tap water for 30 s approximately 10 min prior to saliva collection and will be asked to expectorate into sterile tubes while sitting in an upright position until collecting 3 ml of unstimulated saliva. The quantification of the biomarker in saliva will be assayed using enzyme-linked immunoassay (ELISA).

ELIGIBILITY:
Inclusion Criteria:

* the included participant will be patients smoking cigarette at least 12 months no more than 8 cigarettes per day, patients use electronic vape in categories of low to medium dependance according to the Penn state electronic cigarette dependence index (one time consist of around 15 puffs or last around ten minutes). participants who never consumed tobacco in any form during their lifetime, having minimum of 20 teeth, additionally, all of involved patients having generalized gingivitis with intact periodontium in which they have more than 10% bleeding sites with no PPD >3 mm with no clinical attachment loss according to criteria proposed by (Chapple in,2018).

Exclusion Criteria:

* dual smokers, smokeless tobacco, heavy smokers, patient using high nicotine formula (more than 25 mg/ml), periodontitis patient, patient with systemic diseases, females, participants who had used antibiotics, steroidal or non-steroid anti-inflammatory drugs within the past 6 months, patients who had undergone periodontal therapy within the last 6 months and patients unwilling to participate in study.

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2023-12-20 (Estimated); Primary Completion 2024-03-20 (Estimated); Study Completion 2024-06-20 (Estimated)

PRIMARY OUTCOMES:
the reduction in periodontal parameters | 3 weeks
  (PI,BOP and GI) between the baseline and the endpoints of the study.

SECONDARY OUTCOMES:
the changes between the baseline and 3 weeks for salivary matrix metalloproteinase 8 and 9 concentration. | three weeks

IPD SHARING:
Plan to Share IPD: Undecided